CLINICAL TRIAL: NCT01761760
Title: Game-based Contingency Management for Smoking Cessation
Brief Title: Videogame-based Incentives for Smoking Cessation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There were a number of bugs in the game that meant the participants were not getting the intended intervention.
Sponsor: Rowan University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Bethany Raiff, Assistant Professor, Rowan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5R34DA033536-03 (NIH); R34DA033536 (NIH)
Record Dates: First submitted 2012-12-21; First posted 2013-01-07 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingent (Experimental): Patients will earn game-based incentives contingent on meeting carbon monoxide goals.
  Behavioral: Videogame-based smoking cessation intervention
  Interventions: Behavioral: Videogame-based smoking cessation intervention
- Non-contingent (Active Comparator): Patients will earn game-based incentives independent of meeting carbon monoxide goals.
  Behavioral: Videogame-based smoking cessation intervention
  Interventions: Behavioral: Videogame-based smoking cessation intervention

INTERVENTIONS:
Behavioral: Videogame-based smoking cessation intervention — Patients will enroll in a videogame that is intended to help them quit smoking. They will be given goals for quitting (based on carbon monoxide readings submitted over a secure internet server) and will earn game-based incentives either contingent or noncontingent on meeting those goals.

SUMMARY:
Investigators will be evaluating an online video-game-based smoking cessation intervention that will overcome barriers to treatment such as cost and sustainability. This videogame will be the first of its kind, based on an evidence-based intervention shown to promote smoking abstinence. The findings from this research will be of great public health significance because of the unprecedented reach and relatively low cost, as well as the potential for similar interventions to be developed for other health problems, such as alcohol or drug abuse and medication adherence for chronic illnesses

DETAILED DESCRIPTION:
Cigarette smoking remains the number one cause of preventable morbidity and mortality in the U.S. A number of barriers have been noted that prevent access to smoking cessation interventions, such as lack of clinician training, the time commitment required to implement treatments, and the costs associated with treatment. Thus, it is critically important that more effective interventions be developed, and be made accessible at a relatively low cost, to smokers. We recently developed an Internet-based Contingency Management Intervention (CM),, where participants submit web-camera recorded videos as they exhale into a CO monitor, and they earn money for abstinence. Although the costs associated with providing monetary incentives contingent on smoking abstinence are likely to be less than the costs associated with medical complications caused by smoking, the cost of incentives is often cited as a barrier to CM. Thus, the goals of the present proposal are to markedly decrease costs and increase sustainability of this highly accessible Internet-based CM for smoking cessation.

Using an iterative development process with the help of a team of experts, a social strategy video game intended to be fun and engaging will be developed for Facebook ("Quitters, Incorporated"). Treatment-seeking smokers will be able to earn incentives contingent on meeting web-camera verified CO values consistent with smoking abstinence. Three powerful, evidence-based incentives will be harnessed in this CM. The incentives will consist of: (1) individual contingencies that can be used to improve game play, (2) social contingencies, such as positive feedback and virtual rewards, that can be given to other players to acknowledge their success with abstinence and improve their game play, and (3) group contingencies that will require all members of a group to meet abstinence goals in order to unlock access to certain game features. After game development, we will assess the feasibility, acceptability, enjoyability, and preliminary efficacy of video-game-based CM for smoking cessation. A 7-week pilot study will involve randomly assigning participants (N=100) to either: (1) abstinent contingent, where incentives will be delivered contingent on quitting smoking, or (2) submission contingent, where incentives will be delivered contingent on submitting videos, but independent of quitting smoking.

The outcomes of the pilot study will impact future research in the development of video-game-based CM interventions for smoking, as well as for alcohol and other drug use, and medication compliance in diabetes, asthma, and other conditions. Game-based CM will promote widespread access to this innovative, fun, sustainable intervention at a relatively low cost (the game will be available to play for free), thereby offering the potential to have a substantial public health impact.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* smoking 10+ cigarettes per day
* smoking for 2+ years
* currently wishes to quit smoking
* has a computer at home with Internet access
* U.S. citizen
* literate

Exclusion Criteria:

* smoking other substances (e.g., marijuana, cigars) > 2 times per month
* unstable medical or psychiatric condition that might interfere with the program
* living with someone who smokes in the home
* a job that exposes the person to excessive ambient carbon monoxide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Sustained smoking abstinence | 7 weeks
  Sustained abstinence will be collected via self-report

SECONDARY OUTCOMES:
Self-reports of smoking status, videogame activity, physical and mental health | 7 weeks
  Patients will complete surveys on-line that ask questions regarding smoking status (how many cigarettes smoked per day), videogame activity (how much time is spent playing videogames), psychosocial health (e.g., physical health, mental health).
Carbon monoxide in parts per million collected via a carbon monoxide monitor and submitted over a secure website via a web-camera recorded video. | 7 weeks
  Carbon monoxide will be collected using a carbon monoxide monitor and submitted via. throughout the study to verify smoking abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Raiff, Principal Investigator — Rowan University
Locations (1):
- Rowan University, Glassboro, New Jersey, United States